CLINICAL TRIAL: NCT00091390
Title: Phase II Trial Of Combined High Dose Rate Brachytherapy And External Beam Radiotherapy For Adenocarcinoma Of The Prostate
Brief Title: Radiation Therapy in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0321; CDR0000382120
Record Dates: First submitted 2004-09-07; First posted 2004-09-09 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- External Beam Radiotherapy and High Dose brachytherapy boost (Experimental)
  Interventions: Radiation: High Dose brachytherapy boost; Radiation: External beam radiotherapy

INTERVENTIONS:
Radiation: High Dose brachytherapy boost — 19 Gy in two fractions (on day of placement and 6-24 hours later) before or after external beam radiotherapy, such that all study treatment occurs within 8 weeks.
  Other Names: HDR brachytherapy boost
Radiation: External beam radiotherapy — 45 Gy as 1.8 Gy five days a week for five weeks.
  Other Names: XRT; External beam RT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other sources to damage tumor cells. Internal radiation therapy uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving radiation therapy in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving internal radiation therapy together with external-beam radiation therapy works in treating patients with stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of late grade 3 or greater genitourinary and gastrointestinal toxicity after treatment with external beam radiotherapy and high-dose rate brachytherapy in patients with stage II or III adenocarcinoma of the prostate.

Secondary

* Determine acute grade 3 or greater genitourinary and gastrointestinal toxicity in patients treated with this regimen.
* Determine freedom from biochemical failure in patients treated with this regimen.
* Determine overall survival of patients treated with this regimen.
* Determine disease-specific survival of patients treated with this regimen.
* Determine clinical relapse (local and/or distant) in patients treated with this regimen.
* Develop a quality assurance process for high-dose rate prostate brachytherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to prostate-specific antigen (≤ 10 ng/mL vs 11-20 ng/mL), T stage (T1c-T2c vs T3a-T3b), combined Gleason score (2-6 vs 7 vs 8-10), prior hormonal therapy (no vs yes), and timing of high-dose rate brachytherapy (before external beam radiotherapy vs after external beam radiotherapy).

Patients are followed at 3, 7, 9, and 12 months, every 6 months for 5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, adenocarcinoma of the prostate, clinical stage T1c-T3b, N0, M0.
2. Patient will have clinically negative nodes as established by imaging (pelvic computed tomography (CT), magnetic resonance imaging (MRI)).
3. The patient will be clinically M0.
4. Zubrod status 0-1.
5. No prior pelvic or prostate radiation or chemotherapy for prostate cancer; induction hormonal therapy beginning ≤ 120 days prior to registration is acceptable.
6. One of the following combinations of factors:

   Clinical stage T1c-T2c, Gleason score 2-6 and prostate-specific antigen (PSA) >10 but ≤ 20 Clinical stage T3a-T3b, Gleason score 2-6 and PSA ≤ 20 Clinical stage T1c-T3b, Gleason score 7-10 and PSA ≤ 20
7. Patients must sign a study-specific consent form prior to registration.

Exclusion Criteria:

1. Stage T4 disease.
2. Lymph node involvement (N1).
3. Evidence of distant metastases (M1).
4. Radical surgery for carcinoma of the prostate.
5. Previous hormonal therapy beginning > 120 days prior to registration.
6. Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
7. Prior transurethral resection of the prostate (TURP).
8. Prior invasive malignancy(except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the oral cavity or bladder are permissible).
9. Hip prosthesis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: I-Chow J. Hsu, MD, Study Chair — University of California, San Francisco
Locations (12):
- United States (12):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Cancer Care Consultants Medical Associates at Daniel Freeman Memorial Hospital, Inglewood, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin

REFERENCES:
- [Result] Hsu IC, Bae K, Shinohara K, Pouliot J, Purdy J, Ibbott G, Speight J, Vigneault E, Ivker R, Sandler H. Phase II trial of combined high-dose-rate brachytherapy and external beam radiotherapy for adenocarcinoma of the prostate: preliminary results of RTOG 0321. Int J Radiat Oncol Biol Phys. 2010 Nov 1;78(3):751-8. doi: 10.1016/j.ijrobp.2009.08.048. Epub 2010 Mar 6. PMID 20207506
- [Result] Jacob D, Raben A, Sarkar A, Grimm J, Simpson L. Anatomy-based inverse planning simulated annealing optimization in high-dose-rate prostate brachytherapy: significant dosimetric advantage over other optimization techniques. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):820-7. doi: 10.1016/j.ijrobp.2008.02.009. Epub 2008 May 1. PMID 18455325
- [Derived] Hsu IC, Rodgers JP, Shinohara K, Purdy J, Michalski J, Roach M 3rd, Vigneault E, Ivker RA, Pryzant RM, Kuettel M, Taussky D, Gustafson GS, Raben A, Sandler HM. Long-Term Results of NRG Oncology/RTOG 0321: A Phase II Trial of Combined High Dose Rate Brachytherapy and External Beam Radiation Therapy for Adenocarcinoma of the Prostate. Int J Radiat Oncol Biol Phys. 2021 Jul 1;110(3):700-707. doi: 10.1016/j.ijrobp.2020.11.008. Epub 2020 Nov 10. PMID 33186617

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Started | 129
Eligible and Started Study Treatment | 125
Eligible, Started Treatment, Has AE Data (Eligible, started study treatment, and has adverse event (AE) data) | 115
Completed | 125 (Subjects contributing data to results are considered to have completed the study.)
Not Completed | 4
Not completed — Protocol Violation | 1
Not completed — No protocol treatment | 3

BASELINE CHARACTERISTICS:
Population: Eligible and started protocol treatment
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
Age, Continuous [Median (Full Range); unit: years] | 68 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 99
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 86
  More than one race | 2
  Unknown or Not Reported | 2
Zubrod Performance Scale [Count of Participants; unit: Participants]
  0 (Asymptomatic) | 121
  1 (Symptomatic but completely ambulatory) | 4
Baseline Prostate-Specific Antigen (PSA) [Count of Participants; unit: Participants] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  Participants
    ≤10 | 87
    >10 - ≤20 | 38
Gleason score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    2-6 | 13
    7 | 90
    8-10 | 22
Prior hormone therapy [Count of Participants; unit: Participants] — Did the participant have hormonal therapy within 120 days prior to study registration?
  Participants
    Yes | 54
    No | 71
T Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T1c-T2c | 114
    T3a-T3b | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Late Grade 3-5 Genitourinary (GU) and Gastrointestinal (GI) Adverse Events (AE) at 18 Months
Description: Adverse events (AE) were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. "Late" is defined as occurring after 9 months from the start of study treatment. Because of the lead time of 9 months, the percentage at 18-months was estimated by the 9-month rate using the cumulative incidence method starting at the 10th month. Death was treated as a competing risk.
Time Frame: From 9 to 18 months after start of study treatment
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 2.56 [0.834 to 7.738]
Statistical Analysis 1: Comparison: External Beam Radiotherapy and High Dose Brachytherapy Boost; The study is designed to test whether the 18-month late GU/GI toxicity following the protocol treatment is above 10% (hazard rate of 0.012/month). The sample size is determined so that the probability of rejecting the treatment because of excessive late toxicity is 90% if the true late toxicity rate is 20% (hazard rate of 0.025/month). Ninety-eight patients are required to with an additional 18 months of follow-up to have a statistical power of 90% with one-sided significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Z-test; One-sided; hazard rate = 0.0014, 95% CI 2-sided [0 to 0.003]

2. Secondary Outcome: Number of Participants With Acute Grade 3-5 Genitourinary (GU) and Gastrointestinal (GI) Adverse Events (AE)
Description: Adverse events (AE) were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to AE. Acute is defined as occurring within 9 months from the start of study treatment.
Time Frame: From treatment start to 9 months
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 2.61 [0.100 to 5.95]

3. Secondary Outcome: Percentage of Participants With Biochemical Failure at 10 Years Using American Society for Therapeutic Radiation and Oncology (ASTRO) Definition
Description: The ASTRO criteria for biochemical failure is three consecutive rises in prostate-specific antigen (PSA) level above the nadir after radiation therapy. The PSA nadir is defined as as the lowest PSA value reached immediately before a biochemical failure. The date of failure is midway between the last non-rising PSA and the first rise in PSA. Time to failure is defined as time from registration to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rate is estimated using the cumulative incidence method.
Time Frame: From registration to ten years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 14.7 [8.9 to 21.9]

4. Secondary Outcome: Percentage of Participants With Biochemical Failure at 10 Years Using the Phoenix Definition
Description: The Phoenix criteria for biochemical failure is a rise of 2 ng/mL or more above the nadir after radiation therapy. Time to failure is defined as time from registration to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rate is estimated using the cumulative incidence method.
Time Frame: From registration to ten years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 22.6 [15.3 to 30.6]

5. Secondary Outcome: Percentage of Participants Alive at 10 Years
Description: Overall survival time is defined as time from registration to the date of death from any cause or last known follow-up (censored). Overall survival rate is estimated by the Kaplan-Meier method.
Time Frame: From registration to 10 years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 75.7 [67.2 to 84.1]

6. Secondary Outcome: Percentage of Participants With Death Due to Prostate Cancer at 10 Years
Description: The following will be considered as death due to prostate cancer (failure):
  * Death certified as due to prostate cancer.
  * Death from other causes with active malignancy (clinical or biochemical progression).
  * Death due to complications of treatment, irrespective of the status of malignancy.
  Time to failure is defined as time from registration to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rate is estimated using the cumulative incidence method.
Time Frame: From registration to ten years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 6.4 [2.6 to 12.6]

7. Secondary Outcome: Percentage of Participants With Distant Failure at 10 Years
Description: Distant failure required documentation of regional nodal recurrence or distant disease relapse. Time to failure is defined as time from registration to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rate is estimated using the cumulative incidence method.
Time Frame: From registration to ten years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 7.7 [3.5 to 14.0]

8. Secondary Outcome: Percentage of Participants With Local Failure at 10 Years
Description: Local failure is defined as documented local progression as determined by clinical exam. Time to failure is defined as time from registration to the date of first failure, last known follow-up (censored), or death without failure (competing risk). Failure rate is estimated using the cumulative incidence method.
Time Frame: From registration to ten years
Population: Eligible participants who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | External Beam Radiotherapy and High Dose Brachytherapy Boost
Number analyzed (Participants) | 125
percentage of participants | 1.7 [0.3 to 5.4]

ADVERSE EVENTS:
Groups:
- EBRT and HDR Brachytherapy Boost: External beam radiation therapy (EBRT) and high dose rate (HDR) brachytherapy boost.
Arm/Group | EBRT and HDR Brachytherapy Boost
Serious Adverse Events (participants affected / at risk) | 49/115
Other Adverse Events (participants affected / at risk) | 110/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EBRT and HDR Brachytherapy Boost (N=115)
Hemoglobin (Blood and lymphatic system disorders) | 1
Diarrhea NOS (Gastrointestinal disorders) | 2
Fecal incontinence (Gastrointestinal disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Pain - Other (General disorders) | 1
Infection - Other (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Fanconi syndrome acquired (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 2
Bladder pain (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 21
Renal/genitourinary - Other (Renal and urinary disorders) | 3
Ureteric obstruction (Renal and urinary disorders) | 1
Urethral obstruction (Renal and urinary disorders) | 1
Urethral pain (Renal and urinary disorders) | 6
Urethral stricture (Renal and urinary disorders) | 3
Urinary bladder hemorrhage (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 3
Urogenital hemorrhage (Renal and urinary disorders) | 2
Erectile dysfunction NOS (Reproductive system and breast disorders) | 16
Penile pain (Reproductive system and breast disorders) | 1
Flushing (Vascular disorders) | 1
Hot flushes NOS (Vascular disorders) | 2
Hypertension NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EBRT and HDR Brachytherapy Boost (N=115)
Hemoglobin (Blood and lymphatic system disorders) | 10
Constipation (Gastrointestinal disorders) | 7
Diarrhea NOS (Gastrointestinal disorders) | 30
Proctitis NOS (Gastrointestinal disorders) | 12
Rectal hemorrhage (Gastrointestinal disorders) | 23
Fatigue (General disorders) | 23
Pain - Other (General disorders) | 6
Libido decreased (Psychiatric disorders) | 23
Bladder pain (Renal and urinary disorders) | 10
Cystitis NOS (Renal and urinary disorders) | 11
Pollakiuria (Renal and urinary disorders) | 90
Renal/genitourinary - Other (Renal and urinary disorders) | 21
Urethral obstruction (Renal and urinary disorders) | 9
Urethral pain (Renal and urinary disorders) | 19
Urethral stricture (Renal and urinary disorders) | 7
Urinary incontinence (Renal and urinary disorders) | 24
Urinary retention (Renal and urinary disorders) | 46
Urogenital hemorrhage (Renal and urinary disorders) | 22
Ejaculatory disorder NOS (Reproductive system and breast disorders) | 7
Erectile dysfunction NOS (Reproductive system and breast disorders) | 66
Penile pain (Reproductive system and breast disorders) | 8
Hot flushes NOS (Vascular disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.